CLINICAL TRIAL: NCT06976918
Title: Clinical Research Platform on Treatment, Quality of Life and Outcome of Patients With Primary and Secondary Myelofibrosis and Anemia Who Are JAK Inhibitor Treatment-naïve or JAK Inhibitor Treatment-experienced (RHODOLITE)
Brief Title: Registry Platform Myelofibrosis and Anemia
Acronym: RHODOLITE
Status: Not yet recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: German Study Group for Myeloproliferative Neoplasms (GSG-MPN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: iOM-110507
Record Dates: First submitted 2025-04-29; First posted 2025-05-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Anemia; Myelofibrosis; Anemia; Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis; Anemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the project is to set up a national, prospective, longitudinal, multicenter cohort study, a tumor registry platform, to document uniform data on characteristics, molecular diagnostics, treatment and course of disease and to collect patient-reported outcomes for patients with primary and secondary myelofibrosis and anemia in Germany.

DETAILED DESCRIPTION:
RHODOLITE is a national, prospective, open-label, longitudinal, non-interventional multicenter cohort study (tumour registry platform) to describe treatment in routine clinical practice of myelofibrosis patients in routine care in Germany.

The registry will follow patients for up to three years with the aim to identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments and outcome are documented.

Health-related quality of life (HRQoL) will be evaluated for up to three years.

The RHODOLITE clinical registry is a joint project with the German Study Group for Myeloproliferative Neoplasms (GSG-MPN) and its GSG-MPN Bioregistry (NCT03125707). Details on treatment and outcome will be collected in RHODOLITE clinical registry for up to three years, while long-term follow-up for a minimum of additional five years will be performed in the GSG-MPN Bioregistry.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary or secondary (post-polycythemia vera or post-essential thrombocythemia) myelofibrosis (MF) (Note: diagnosis according to WHO-2017, ICC-2022 or WHO-2022 or IWG-MRT criteria, respectively).
* Diagnosis of anemia at the time of enrollment as per individual, clinical assessment by the local physician.
* Start of first or subsequent systemic treatment for MF.
* Informed consent and registration for the GSG-MPN Bioregistry.
* Willingness and capability to participate in PRO assessment.
* Signed and dated informed consent form for RHODOLITE at the latest six weeks after start of the respective systemic MF treatment.

Exclusion Criteria:

* No systemic therapy for diagnosed primary or secondary MF.
* Planned allogenic stem cell transplantation (allo-SCT) or active participation in an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with primary myelofibrosis or post-polycythemia vera or post-essential thrombocythemia myelofibrosis (MF) with anemia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Documentation of systemic treatment for MF and therapy sequences | 3 years per patient
  Types and frequencies of systemic treatment for MF during observation time.

SECONDARY OUTCOMES:
Hematologic response | 3 years per patient
  Frequencies of hematologic response (improved, stable, worsened) per line of treatment
Splenic response | 3 years per patient
  Frequencies of splenic response (improved, stable, worsened) per line of treatment
Overall response rate (ORR) | 3 years per patient
  Documentation of ORR per line of treatment
Progression free survival (PFS) | 3 years per patient
  Documentation of PFS per line of treatment
Overall survival | 3 years per patient
  Documentation of OS per line of treatment
Health-related quality of life (Patient-reported outcome, PRO) | 3 years per patient
  European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (EORTC QLQ-C30, the lower the score the better the QoL)
Assessment of Myelofibrosis-related symptoms | 3 years per patient
  Myelofibrosis Symptom Assessment form (MFSAF) questionnaire 7-day Recall

CONTACTS AND LOCATIONS:
Overall Officials: Konstanze Döhner, Prof. Dr. med., Study Chair — University Hospital Ulm, Germany; Steffen Koschmieder, Prof. Dr. med., Study Chair — University Hospital Aachen, Germany
Locations (1):
- Multiple sites all over Germany, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No